CLINICAL TRIAL: NCT05984511
Title: TACE Plus Atezolizumab/Bevacizumab and I-125 Seeds Brachytherapy for HCC With Branch PVTT: A Phase III, Randomized Clinical Trial
Brief Title: TACE Plus Atezolizumab/Bevacizumab and I-125 Seeds Brachytherapy for HCC With Branch PVTT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University Cancer Center (SUSUCC) (Unknown); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Maoming People's Hospital (Other); Shandong Province Third hospital (Other)
Responsible Party: Principal Investigator, Huang Mingsheng, The director of Department of Interventional Radiology, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: II2023-162-02
Record Dates: First submitted 2023-07-26; First posted 2023-08-09 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma; Hepatic Portal Vein Tumor Invasion; Tumor Thrombus
Keywords: Hepatocellular Carcinoma (HCC); Portal vein tumor thrombosis (PVTT); Transcatheter arterial chemoembolization (TACE); I-125 Seeds Brachytherapy; Atezolizumab plus Bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label trial, randomized controlled trial to evaluate the efficacy and safety of TACE-AB-I compared with TACE-AB for the treatment of HCC with branch PVTT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TACE plus Atezolizumab/Bevacizumab and I-125 Seeds Brachytherapy (TACE-AB-I) (Experimental): TACE will be performed for the patients after randomization. Iodion-125 seeds will be implanted into the PVTT under CT guidance within 3-7 days after the first TACE.
  Atezolizumab/bevacizumab (1,200 mg atezolizumab plus 15 mg/kg bevacizumab intravenously every 3 weeks) will be started at 3-7 days after the first TACE and I-125 Seeds Brachytherapy.
  TACE and iodion-125 seeds implantation can be repeated on demand during follow-up based on the evaluation of laboratory and imaging examination.
  Interventions: Procedure: I-125 Seeds Brachytherapy in PVTT; Procedure: Transcatheter arterial chemoembolization; Drug: Atezolizumab plus Bevacizumab
- TACE and Atezolizumab/Bevacizumab (TACE-AB) (Active Comparator): TACE will be performed for the patients after randomization. Atezolizumab/bevacizumab (1,200 mg atezolizumab plus 15 mg/kg bevacizumab intravenously every 3 weeks) will be started at 3-7 days after the first TACE.
  TACE can be repeated on demand during follow-up based on the evaluation of laboratory and imaging examination.
  Interventions: Procedure: Transcatheter arterial chemoembolization; Drug: Atezolizumab plus Bevacizumab

INTERVENTIONS:
Procedure: I-125 Seeds Brachytherapy in PVTT — Iodine125 seed implantation into the PVTT was conducted 3-7 days after TACE when the results of the liver function tests were comparable to those obtained before TACE. Pre-procedural planning was conducted using a three-dimensional conformal radiation therapy treatment planning system (TPS) to determine the number of Iodine125 seeds required, the target location for implantation, the best percutaneous puncture site and the access route. The targeted zone for implantation was the tumour thrombosis in the segmental portal vein, left/right portal vein. Implantation was guided by CT, and the Iodine125 seeds were implanted into the PVTT using 18 G needles and the implantation gun that housed the Iodine125 seeds in the cartridge chamber.
  Other Names: Iodine-125 Seeds Implantation
  Arms: TACE plus Atezolizumab/Bevacizumab and I-125 Seeds Brachytherapy (TACE-AB-I)
Procedure: Transcatheter arterial chemoembolization — TACE: cTACE (conventional TACE) or dTACE (drug-eluting beads TACE).
  Other Names: TACE
Drug: Atezolizumab plus Bevacizumab — Atezolizumab/bevacizumab (1,200 mg atezolizumab plus 15 mg/kg bevacizumab intravenously every 3 weeks) .
  Other Names: atezolizumab-bevacizumab; Atez/Bev treatment

SUMMARY:
The present study aimed to assess the effectiveness of the combination treatment of Atezolizumab/Bevacizumab, transcatheter arterial chemoembolization (TACE) and I-125 Seeds Brachytherapy (TACE-AB-I) in patients with advanced hepatocellular carcinoma (HCC) and portal vein tumor thrombosis (PVTT). The investigators confirmed that the combination therapy yielded better survival data than the combined administration of Atezolizumab/Bevacizumab and TACE (TACE-AB) in patients with advanced HCC and Type I/II PVTT (Based on Cheng's PVTT classification).

DETAILED DESCRIPTION:
This is a multicenter, open-label trial, randomized controlled to evaluate the efficacy and safety of TACE-AB-I compared with TACE-AB for the treatment of HCC with branch PVTT. 234 HCC patients with branch PVTT will be enrolled in this study. The Patients will be treated with TACE-AB-I or TACE-AB using a 1:1 randomization scheme. TACE will be performed for the patients after randomization. Atezolizumab/bevacizumab (1,200 mg atezolizumab plus 15 mg/kg bevacizumab intravenously every 3 weeks) will be started at 3-7 days after the first TACE and I-125 Seeds Brachytherapy and last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. For patients in the TACE-AB-I arm, iodion-125 seeds will be implanted into the PVTT (according to the pre-operative planning) under CT guidance within 3-7 days after the first TACE. TACE and iodion-125 seeds implantation can be repeated on demand during follow-up based on the evaluation of laboratory and imaging examination.

ELIGIBILITY:
Inclusion Criteria:

* Age between18 and 75 years;
* Has a diagnosis of HCC confirmed by radiology, histology, or cytology;
* Type I PVTT or type II PVTT;
* Child-Pugh class A;
* Eastern Cooperative Group performance status (ECOG) score of 0-1;
* No prior systemic therapy for HCC.
* Adequate hematologic and end-organ function;
* At least one measurable intrahepatic target lesion.

Exclusion Criteria:

* Diffuse HCC;
* Cholangiocarcinoma, fibrolamellar, sarcomatoid hepatocellular carcinoma, and mixed hepatocellular/cholangiocarcinoma subtypes (confirmed by histology, or pathology) are not eligible;
* Evidence of extrahepatic spread (EHS);
* Any condition representing a contraindication to TACE or I-125 seeds brachytherapy as determined by the investigators;
* Evidence or history of bleeding diathesis or any hemorrhage or bleeding event >CTCAE grade 3 within 4 weeks prior to randomization;
* Active or history of autoimmune disease or immune deficiency;
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding;
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment;
* Evidence of bleeding diathesis or significant coagulopathy;
* Pregnant or breastfeeding females;
* Significant cardiovascular disease;
* Severe infection, such as active tuberculosis;
* Serious medical comorbidities;
* History of organ or cells transplantation;
* History of other uncurable malignancies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years
  Time from randomization to death from any cause.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Time from randomization to disease progression (mRECIST) or death from any cause, whichever occurred first.
Objective response rate (ORR) | 2 years
  The percentage of patients who had a best overall tumor response rating of CR and PR (mRECIST).
Duration of portal patency | 2 years
  The time from randomization until the date that complete portal vein occlusion was confirmed (if the portal vein is patent at diagnosis).
Adverse events (AEs) | 2 years
  Number of patients with AE, treatment-related AE (TRAE), AE of special interest (AESI), serious adverse event (SAE), assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Mingsheng Huang, M.D. & Ph.D., Principal Investigator — Department of Interventional Radiology, The Third Affiliated Hospital of Sun Yat-sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No
Plan to share IPD with collaborators.